CLINICAL TRIAL: NCT02675920
Title: A Prospective Cohort Study to Compare Contrast Enhanced Liver CT and Ultrasonography for Hepatocellular Carcinoma Surveillance in High-risk Group of HCC: Preliminary Study
Brief Title: A Study of HCC High Risk Group Using Two Surveillance Tools
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Taejoon Pharmaceutical Co., Ltd. (Industry); Reyon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH-2013-2284
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: HCC
Keywords: surveillance; ultrasonography; computed tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- High risk group of HCC: known high risk group of HCC according to AASLD guideline. And patients whose risk index is equal to or higher than 2.33.
  Risk Index = 1.65 (if the prothrombin activity is <=75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <=100x10(3)/mm3) + 0.74 (if the presence of anti-hepatitis C virus [HCV] or hepatitis B surface antigen [HBsAg] is positive).
  Patients undergo ultrasonography and LDCT using non-ionic monomer iodinated CT contrast media biannually and the interval between ultrasound and LDCT is within 30 days.
  Interventions: Drug: non-ionic monomer iodinated CT contrast media

INTERVENTIONS:
Drug: non-ionic monomer iodinated CT contrast media — patients underwent contrast-enhanced CT using aforementioned CT contrast media (non-ionic monomer iodinated CT contrast media)
  Other Names: contrast enhanced CT

SUMMARY:
The purpose of this study is to compare sensitivity for hepatocellular carcinoma (HCC) of bi-annual ultrasonography and low dose computed tomography (LDCT) in patients at high risk of HCC.

DETAILED DESCRIPTION:
Patients at high risk of HCC are recommended to undergo biannual surveillance using ultrasound. In this study, LDCT is performed in addition to biannual ultrasound surveillance in eligible patients to compare their sensitivity for HCC. Standard of reference would be follow-up imaging and/or gadoxetic acid-enhanced liver MRI.

ELIGIBILITY:
Inclusion Criteria:

All conditions have to be satisfied to be enrolled.

* > 20 years
* high risk group of HCC according to AASLD guideline
* risk index > = 2.33
* currently on regular biannual surveillance using ultrasonography
* sign informed consent

Exclusion Criteria:

Patients with any of following condition cannot be enrolled.

* previously diagnosed with HCC
* any contraindication of contrast enhanced CT including allergic reaction to iodine
* history of other malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk of HCC AND High Risk Index (>=2.33)
  Risk Index = 1.65 (if the prothrombin activity is <=75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <=100x10(3)/mm3) + 0.74 (if the presence of anti-hepatitis C virus [HCV] or hepatitis B surface antigen [HBsAg] is positive).
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Detection rate of patients with HCC | 18 months
  from the 1st LDCT/US screening to six months follow-up after last (12 months after 1st LDCT/US) LDCT/US screening

SECONDARY OUTCOMES:
Detection rate of patients with early HCC | 18 months
  from the 1st LDCT/US screening to six months follow-up after last (12 months after 1st LDCT/US) LDCT/US screening
False referral rate | 18 months
  from the 1st LDCT/US screening to six months follow-up after last (12 month after 1st LDCT/US) LDCT/US screening

OTHER OUTCOMES:
radiation dose per patient | 12 months
  from the 1st LDCT/US screening to last LDCT/US screening

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No